CLINICAL TRIAL: NCT01265134
Title: Efficacy of Arch Insoles in the Dynamic Postural Control for the Elderly
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Chi-Hsien Chen, Department of Physical Medicine & Rehabilitation, Taipei Medical University- Wan fang Hospital
Other Study IDs: 99063
Record Dates: First submitted 2010-12-21; First posted 2010-12-22 (Estimated); Last update posted 2011-01-03 (Estimated); Status verified 2010-12

CONDITIONS: Balance; Distorted
Keywords: the elders; falling; loss balance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Experimental Group: the healthy elders
- Control Group: the elders who have fallen once

SUMMARY:
The purpose of this study is to measure the ability of balance controlling and test the evaluation of clinical trials with different arch insoles. The investigators want to find out the difference and efficacy of arch insoles in the dynamic postural control for the elderly.

ELIGIBILITY:
Inclusion Criteria:

* no cognition problem. (mini-mental state examination [MMSE] > 23)
* no sensory or motor problem
* no use drugs about balance control
* lower extremity without any traumatic injury

Exclusion Criteria:

* Cognition impairment
* with specific neurological deficits resulting from neuropathy, neuromuscular disorders or spinal stenosis
* use drugs about balance control
* total joint arthroplasty

Ages: 65 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: the elders
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2010-10; Study Completion 2011-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Hsien Chen, Principal Investigator — Taipei Medical University WanFang Hospital
Locations (1):
- Taipei Medical University - Wanfang Hospital, Taipei, Taiwan